CLINICAL TRIAL: NCT04076865
Title: A Mechanistic Evaluation of the Nociceptive Desensitization Induced by Repeated Administration of Topical Local Anaesthetic Mixture of Lidocaine and Prilocaine (EMLA) in a Model of Histaminergic and Non-histaminergic Itch.
Brief Title: Evaluation of the Effect Induced by Repeated Administration of Topical Local Anaesthetic (EMLA) on Itch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, Principal Investigator, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-20190043
Record Dates: First submitted 2019-08-30; First posted 2019-09-03 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Lidocaine; Itch
MeSH Terms: conditions — Pruritus | interventions — Lidocaine, Prilocaine Drug Combination; Lidocaine; UBE3A protein, human; Histamine

STUDY DESIGN:
Masking Description: The participant are blind about the location of EMLA and placebo application
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EMLA (Experimental)
  Interventions: Drug: EMLA (lidocaine) +Itch (Histamine and cowhage)

INTERVENTIONS:
Drug: EMLA (lidocaine) +Itch (Histamine and cowhage) — Cutaneous anaesthesia: will be topically induced by using EMLA cream 5%, a local anaesthetic cream consisting of equal parts of lidocaine and prilocaine (1g contains 25 mg of lidocaine and 25 mg of prilocaine, AstraZeneca A/S, Albertslund, Denmark).
  Histamine: To deliver histamine, standard allergy skin prick test (SPT) lancets are applied.
  Cowhage: Cowhage spicules are 1-2 mm in length and have diameter of 1-3 um at their tip, once inserted into the epidermis, the spicules evoke a moderate sensation of itch and to a lesser extent sensations of burning and stinging pain.

SUMMARY:
In this experiment, the investigators would like to study if the repeated application of local cuaneous anaesthetic EMLA cream will reduce itch induced by small needles from the plant mucuna pruriens (also known as cowhage) and histamine (an itch proving substance formed in the body).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids or other drugs
* Previous or current neurologic, musculoskeletal or mental illnesses
* Lack of ability to cooperate
* Current use of medications that may affect the trial
* Skin diseases
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Acute or chronic pain
* Participation in other trials within 1 week of study entry (4 weeks in the case of pharmaceutical trials)
* Known history of anaphylactic shock, or local allergy (contact dermatitis) to lidocaine, prilocaine or other local anaesthetics of the amide type.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Superficial blood perfusion | Change from baseline, up to three days after the first session
  is measured by a Speckle contrast imager (FLPI, Moor Instruments, England).
Warm Detection Thresholds and Heat Pain Thresholds | Change from baseline, up to three days after the first session
  The tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Pain to Supra-threshold Heat Stimuli | Change from baseline, up to three days after the first session
  The tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Alloknesis | Change from baseline, up to three days after the first session
  Alloknesis is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 miliNewton of force).
Mechanical Pain Thresholds and Sensitivity | Change from baseline, up to three days after the first session
  This test is performed using a pin-prick set (Aalborg University, Aalborg). The set consists of 8 needles each having a diameter of 0.6 mm and different force applications: 0.8, 1.6, 3.2, 6.4, 12.8, 25.6, 50.1 and 60.0 g
Pain rating | only on day 3 (third session)
  The subject will rate the pain for 9 min by using a a visual analog scale (VAS) on a tablet. This scale goes from 0 to 100. 0 indicates 'no pain' and 100 indicates 'worst imaginable pain'.

SECONDARY OUTCOMES:
Itch rating | only on day 3 (third session)
  The subject will rate the itch for 9 min by using a a visual analog scale (VAS) on a tablet. This scale goes from 0 to 100. 0 indicates 'no itch' and 100 indicated 'worst imaginable itch'.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Lo Vecchio, Principal Investigator — Aalborg University
Locations (1):
- Aalborg University, Aalborg, North Denmark, Denmark